CLINICAL TRIAL: NCT03052049
Title: Prostatic Artery Embolization (PAE) for Treatment of Signs and Symptoms of Benign Prostatic Hyperplasia (BPH)
Brief Title: Prostatic Artery Embolization (PAE) for Treatment of Signs and Symptoms of Benign Prostatic Hyperplasia (BPH) Using Bead Block Microspheres
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: BTG International Inc. (Other)
Responsible Party: Principal Investigator, Riad Salem, Professor of Radiology, Medicine and Surgery; Chief, Vascular and Interventional Radiology, Northwestern University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STU 00204385
Record Dates: First submitted 2017-02-08; First posted 2017-02-14 (Actual); Results first posted 2023-04-12 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2023-10

CONDITIONS: Benign Prostatic Hyperplasia (BPH)
Keywords: Prostate Artery Embolization
MeSH Terms: conditions — Prostatic Hyperplasia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Prostate Artery Embolization (Experimental): There is only one arm of this study where patients receive Prostate Artery Embolization
  Interventions: Device: Prostate Artery Embolization

INTERVENTIONS:
Device: Prostate Artery Embolization — The PAE procedure will be completed on all enrolled patients in Interventional Radiology includes a pelvic/prostate angiogram and embolization with Bead Block microspheres to slow/block blood flow to the prostate.
  Other Names: The interventional type is a procedure

SUMMARY:
This is an open-labeled, non-randomized feasibility study to evaluate the safety of prostate artery embolization (PAE) for the treatment of lower urinary tract symptoms attributed to benign prostatic hyperplasia (BPH).

DETAILED DESCRIPTION:
This pilot study will be a single center, open labeled, non-randomized feasibility study to evaluate the initial safety of PAE for the treatment of symptomatic bladder outlet obstruction. 30 adult male subjects will be enrolled in this study. If eligible patients will undergo the prostate artery embolization procedure in the Interventional Radiology department. An angiogram of the prostate arteries will be done. Small beads called Bead Block microspheres will be injected into the prostate artery to slow blood flow to the prostate in the hope of providing relief with minimal side effects and complications, for lower urinary tract symptoms caused by BPH. After the procedure the patient will be followed at 4 weeks, 12 weeks, 6 months, and 12 months post procedure.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of LUTS secondary to BPH refractory to/contraindicated for medical treatment. Patients with indwelling foley catheters will be treated with culture directed antibiotics one time for 5-7 days. The catheter will be removed so urodynamic testing and cystoscopy can be completed as part of the screening visit. It will be replaced when testing is completed.
* Ability to understand and the willingness to sign a written informed consent.
* Prostate volumes 40 - 200 gm. May include 30-39 gm if the subject has a long history of ineffective response to combination medical treatments (alpha-blocker and a 5-alpha reductase inhibitor) for at least 6 months.
* Men ≥ 45 years of age
* IPSS symptom score ≥ 18 and IPSS bother score ≥ 3
* Peak flow rate Qmax≤ 12 with voided volume ≥125 cc
* For men 45-59 years old: Prostate Specific Antigen) PSA < 2.5 (or) PSA 2.5-20 with a documented negative biopsy within previous 12 months.
* For men >60: PSA < 4 (or) PSA 4-20 with a documented negative biopsy within previous 12 months.

Exclusion Criteria:

* History of prostate or bladder cancer, pelvic radiation, untreated bladder stones,
* On alpha-blockers within the past 2 weeks unless on a stable dose of medication with a stable urination pattern for 2 weeks prior to enrollment and the willingness to stay on the same dose for the duration of the study or if criteria are met at the 1 year follow up visit and/or part of a Trial without catheter (TWOC) and patient is currently in Acute Urinary Retention (AUR).
* On 5-alpha reductase inhibitors within the past 6 months. Unless on a stable dose of medication with a stable urination pattern for 30 days prior to enrollment and the willingness to stay on the same dose for the duration of the study or if criteria are met at the 1 year follow up visit
* On phenylephrine, pseudoephedrine, imipramine, an anticholinergic or cholinergic medication within the past 2 weeks. Unless on a stable dose of medication with a stable urination pattern for 2 weeks prior to enrollment and the willingness to stay on the same dose for the duration of the study or if criteria are met at the 1 year follow up visit.
* On estrogen, androgen, any drug producing androgen suppression, or anabolic steroids within the past 4 months unless on stable dose of medication for 30 days prior to enrollment and the willingness to stay on the same dose for the duration of the study or if criteria are met at the 1 year follow up visit
* Daily use of a pad or device for incontinence required.
* Current urethral strictures/Bladder neck contracture (BNC) (past urethral strictures which have been treated successfully > 6 months prior are eligible)
* renal insufficiency (i.e. creatinine > 1.8)
* Known primary neurologic conditions such as multiple sclerosis or Parkinson's disease or other neurological diseases known to affect bladder function.
* Neurogenic bladder, Hypotonic Bladder
* Prior treatment for urinary incontinence
* Penile prosthesis.
* Artificial urinary sphincter.
* Documented bacterial prostatitis within the past year.
* Active urinary tract infection (UTI) unless in case of regular catheter dependence and thought to represent colonization.
* History of chronic prostatitis within the last 1 year
* Known bleeding disorders (e.g. VWD)
* Prior prostate procedures (e.g. Transurethral Microwave Therapy (TUMT), Transurethral Needle Ablation of the Prostate (TUNA), Water-induced Thermotherapy (WIT), Transurethral Resection of the Prostate (TURP), Photoselective Vaporization of the Prostate (PVP)
* Prior treatment for overactive bladder (e.g. intravesical botox)
* Enrolled in another treatment trial for any disease within the past 30 days
* Declines or unable to provide informed consent
* Condition precluding catheter-based intervention (ie occluded vessel, severe atheromatous disease)
* Any serious medical condition likely to impede successful completion of the study, such as certain mental disorders, uncontrolled diabetes, cardiac arrhythmias, cardiac disease including congestive heart failure, significant respiratory disease, or known immunosuppression.
* A history of rectal malignancy
* Prior surgical prostate intervention
* Interest in future fertility
* Allergy to iodinated contrast agents not responsive to steroid premedication regimen
* Contraindication to conscious sedation

Min Age: 45 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2017-09-06 (Actual); Primary Completion 2022-09-26 (Actual); Study Completion 2022-09-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Riad Salem, MD, Principal Investigator — Northwestern University; Matthias Hofer, MD, Study Chair — Northwestern University; Bartley Thornburg, MD, Study Chair — Northwestern University; Kush Desai, MD, Study Chair — Northwestern University; Ahsun Riaz, MD, Study Chair — Northwestern University; Samdeep Mouli, MD, Study Chair — Northwestern University
Locations (1):
- Northwestern, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from both the Interventional Radiology and urology clinics at Northwestern Memorial Hospital in Chicago IL between 2017- 2022.
Period: Overall Study
Arm/Group | Prostate Artery Embolization
Started | 28 (28 subjects were enrolled between October 2017 and January 2020.)
Completed | 26 (26 subjects were treated and 2 withdrew before treatment.)
Not Completed | 2
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Arm/Group | Prostate Artery Embolization
Number analyzed (Participants) | 26
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 12
  >=65 years | 14
Age, Continuous [Mean (Full Range); unit: years] | 66 [52 to 78]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 26
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 25
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 23
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 26
Urinary Retention Requiring an Indwelling Catheter [Count of Participants; unit: Participants] | 1
Length of BPH symptoms (years) [Mean (Full Range); unit: years] | 6 [0.5 to 20]
Total Prostate Volume [Mean (Full Range); unit: cm^3] — Prostate volume was obtained from MRI imaging of the prostate and reported in cm^3.
  cm^3 | 81.0 [26.1 to 196.0]
Blood urea Nitrogen (BUN) [Mean (Full Range); unit: mg/dl] | 17.5 [8.0 to 41]
Creatinine (mg/dl) [Mean (Full Range); unit: mg/dl] | 1.0 [0.6 to 1.71]
International Normalized ratio (INR) [Mean (Full Range); unit: ratio] — International Normalized Ratio (INR) resulted as a ratio.
  ratio | 1.0 [0.9 to 1.20]
PSA (ng/ml) [Mean (Full Range); unit: ng/ml] | 4.6 [0.2 to 17.4]
percentage of Free PSA [Mean (Full Range); unit: percentage] — % Free PSA is the amount of the protein prostate-specific antigen (PSA) in the blood that is not attached to other proteins. It is compared with the amount of PSA in the blood that is attached to other proteins. The amount of free PSA is higher in men with benign prostatic hyperplasia (BPH).
  percentage | 21.0 [9.2 to 27.0]
% Subjects with Abnormal Screening Urinalysis (RBCs) >4 per high Power Field [Number; unit: percentage] | 88
% Subjects with Abnormal Screening Urinalysis (WBCs) >5 per high Power Field [Number; unit: percentage] | 65

OUTCOME MEASURES:

1. Primary Outcome: Number of Reported Treatment-related Adverse Events (AE) as Assessed by NCI CTCAE Grading Scale .
Description: The number of graded adverse events was recorded to evaluate safety. They were graded using the following scale at 1, 3, 6, and 12 months post procedure:
  Mild (grade 1): the event causes discomfort without disruption of normal daily activities Moderate (grade 2): the event causes discomfort that affects normal daily activities Severe (grade 3): the event makes the patient unable to perform normal daily activities or significantly affects his/her clinical status Life-threatening (grade 4): the patient was at risk of death at the time of the event Fatal (grade 5): the event caused death.
Time Frame: 1 year
Population: Events
Measure: Number; unit: events
Arm/Group | Prostate Artery Embolization
Number analyzed (Participants) | 26
events
  Grade 1 AE Mild | 6
  Grade 2 AE Moderate | 10
  Grade 3 AE Severe | 0
  Grade 4 AE life threatening | 0
  Grade 5 AE Fatal | 0
Statistical Analysis 1: Comparison: Prostate Artery Embolization; Test type: Other — t-test; p = 0.05, t-test, 2 sided — P value was calculated with threshold of significance <0.05; p value = 0.05 — P value was calculated with threshold of significance <0.05

2. Secondary Outcome: Change in International Prostate Symptom Score (IPSS)
Description: Questionnaire- IPSS has 7 questions. Answer choices are as follows. The International Prostate Symptom Score (IPSS) can be utilized to measure the severity of lower urinary tract symptoms.
  It is a validated, reproducible scoring system to assess disease severity and response to therapy.
  The IPSS is made up of 7 questions related to voiding symptoms. Scores can range from 0-35 with 0 being the better outcome and 35 the worst outcome.
  Question 1-6 0-Not at all
  1. Less than 1 time in 5
  2. Less than half the time
  3. About half the time
  4. More than half the time
  5. Almost always
  Question 7 0-None 1-1 time 2-2 times 3-3 times 4-4 times 5-5 or more times
Time Frame: Baseline, 1, 3, 6, 12 months post procedure
Population: Not all participants completed the questionnaire at all time points.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Prostate Artery Embolization
Number analyzed (Participants) | 26
score on a scale
  Baseline | 25 (5.2)
  1 month follow up: number analyzed (Participants) | 22
  1 month follow up | 13 (5.4)
  3 month follow up: number analyzed (Participants) | 23
  3 month follow up | 8 (5.6)
  6 month follow up: number analyzed (Participants) | 21
  6 month follow up | 7 (6.3)
  12 month follow up: number analyzed (Participants) | 21
  12 month follow up | 9 (7.3)
Statistical Analysis 1: Comparison: Prostate Artery Embolization; Test type: Other; p = 0.05, t-test, 2 sided — P value was calculated and a value of <0.05 was considered significant

3. Secondary Outcome: Change in Quality of Life (QOL) Bother Score
Description: The total score ranges from 0-6 with 0 being the best outcome and 6 being the worst outcome.
  Questionnaire- answers choices are as follows:
  0- Delighted
  1. Pleased
  2. Mostly Satisfied
  3. Mixed about equality satisfied and dissatisfied
  4. Mostly Dissatisfied
  5. Unhappy
  6. Terrible
Time Frame: Baseline, 1, 3, 6, 12 months post procedure
Population: Not all participants completed this score at all data points.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Prostate Artery Embolization
Number analyzed (Participants) | 26
score on a scale
  Baseline | 5 (0.9)
  1 month follow up: number analyzed (Participants) | 23
  1 month follow up | 2 (1.4)
  3 month follow up: number analyzed (Participants) | 24
  3 month follow up | 1 (1.7)
  6 month follow up: number analyzed (Participants) | 22
  6 month follow up | 1 (1.8)
  12 month follow up: number analyzed (Participants) | 22
  12 month follow up | 1 (1.6)
Statistical Analysis 1: Comparison: Prostate Artery Embolization; Test type: Other; p = 0.05, t-test, 2 sided — P value was calculated and a value of <0.05 was considered significant

4. Secondary Outcome: Change in Benign Prostatic Hyperplasia (BPH) Impact Index Score
Description: The BPH Impact Index is to assess the impact of BPH symptoms on patient health and functioning. It is a self-administered questionnaire with 4 questions about urinary problems during the past month regarding physical discomfort, worry about health, how bothersome symptoms are, and whether the symptoms are interfering with doing usual activities.The BII is an evaluative index useful in measuring the magnitude of change in the impact of BPH-LUTS within a person over time.
  Scores range from 0-13 with 0 being the best outcome and 13 being the worst.
  Questionnaire- consists of 4 questions; answer choices are as follows Question 1: 0-none, 1-only a little, 2-some, 3-a lot Question 2: 0-none, 1-only a little, 2-some, 3-a lot Question 3: 0-not at all bothersome, 1- bothers me a little, 2-bothers me some, 3-bothers me a lot Question 4: 0-none of the time, 1- a little of the time, 2- some of the time, 3-most of the time, 4-all of the time
Time Frame: Baseline, 1, 3, 6, 12 months post procedure
Population: Not all participants answered this questionnaire at all data points.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Prostate Artery Embolization
Number analyzed (Participants) | 26
score on a scale
  Baseline | 9 (2.2)
  1 month follow up: number analyzed (Participants) | 25
  1 month follow up | 3.5 (2.7)
  3 month follow up | 2.5 (2.9)
  6 month follow up: number analyzed (Participants) | 25
  6 month follow up | 2.3 (3.1)
  12 month follow up: number analyzed (Participants) | 22
  12 month follow up | 2.1 (2.4)
Statistical Analysis 1: Comparison: Prostate Artery Embolization; Test type: Other; p = 0.05, t-test, 2 sided — P value was calculated and a value of <0.05 was considered significant

5. Secondary Outcome: Change in Peak Urine Flow (Qmax)
Description: Peak Urine Flow (Qmax) from urodynamic assessments will be summarized comparing baseline to follow up measurements
Time Frame: Baseline, 1, 3, 6, and 12 months post procedure
Population: Low numbers of participants for the 6 month and 12 month follow up visits are attributed to COVID when no visits were being made in person.
Measure: Mean (Standard Deviation); unit: ml/second
Arm/Group | Prostate Artery Embolization
Number analyzed (Participants) | 26
ml/second
  baseline | 5.9 (3.4)
  1 month follow up: number analyzed (Participants) | 20
  1 month follow up | 9.9 (9.1)
  3 month follow up: number analyzed (Participants) | 21
  3 month follow up | 13.2 (13.9)
  6 month follow up: number analyzed (Participants) | 2
  6 month follow up | 7 (0.8)
  12 month follow up: number analyzed (Participants) | 11
  12 month follow up | 9.1 (5.2)
Statistical Analysis 1: Comparison: Prostate Artery Embolization; Test type: Superiority; p = 0.05, t-test, 2 sided — P value was calculated and a value of <0.05 was considered significant

ADVERSE EVENTS:
Time Frame: Adverse events were evaluate at each follow up visit at 1 month, 3 months, 6 months and 12 months after the procedure for each subject. Each subject was evaluated over the study duration on average 1 year or 12 months.
Arm/Group | Prostate Artery Embolization
All-Cause Mortality (participants affected / at risk) | 0/26
Serious Adverse Events (participants affected / at risk) | 0/26
Other Adverse Events (participants affected / at risk) | 10/26
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Prostate Artery Embolization (N=26)
Renal and Urinary Adverse Events (Renal and urinary disorders) | 10 (16) — Events associated with urinary tract or genital region, damage to bladder floor, trigone, sphincters, rectum, incontinence, infections, secondary surgical interventions, transient post procedure events, deaths

LIMITATIONS AND CAVEATS:
We were funded for 30 procedures and anticipated 30 patients. 2 of the patients needed a second procedure, resulting in 28 patients enrolled.

Also, during COVID, there were patients that did not come for Qmax testing.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-11-19): https://cdn.clinicaltrials.gov/large-docs/49/NCT03052049/Prot_SAP_000.pdf